CLINICAL TRIAL: NCT06063096
Title: Gastrointestinal Tolerance of D-allulose in Children: an Acute, Randomised, Double-blind, Placebo-controlled, Cross-over Study
Brief Title: Gastrointestinal Tolerance of D-allulose in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tate & Lyle (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TateLyle
Record Dates: First submitted 2023-08-02; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Acute, randomised, double-blind, placebo-controlled, cross-over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allulose Dose 1 (Active Comparator): Fruit-flavoured drink with allulose at Dose 1 (2.5 g per 120 ml)
  Interventions: Dietary Supplement: D-allulose
- Allulose Dose 2 (Active Comparator): Fruit-flavoured drink with allulose at Dose 2 (4.3 g per 120 ml)
  Interventions: Dietary Supplement: D-allulose
- Placebo Comparator: Control (CON) (Placebo Comparator): Control drink containing high fructose corn syrup.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-allulose — Fruit-flavoured drink with d-allulose at 2 dosages
  Arms: Allulose Dose 1; Allulose Dose 2
Dietary Supplement: Placebo — Fruit-flavoured drink with high fructose corn syrup
  Arms: Placebo Comparator: Control (CON)

SUMMARY:
D-allulose, a low-calorie sugar, provides an attractive alternative to sucrose and added sugars in products. This study aimed to verify the tolerance of d-allulose in children, in doses that are Generally Recognised As Safe (GRAS) and below maximum tolerable levels on g/kg basis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children of 6 to 8 years of age
2. Weight-for-age between the 5th and the 90th percentile as per the Centre for Disease Control and Prevention Growth Charts
3. Accustomed to having lunch between 12.00 pm and 2.30 pm
4. Routinely had up to 3 bowel movements per day or as few as 3 bowel movements per week
5. Were able to drink 120 ml within 30 minutes
6. With parents willing to continue their child's normal food and beverage intake and physical activity throughout the duration of the study
7. With parents willing and able to attend for all 7 visits

Exclusion Criteria:

1. Any major trauma or surgical event within the 3 months prior to screening
2. History or presence of clinically significant endocrine or GI disorder
3. Functional GI Disorders in accordance with Rome III Diagnostic Questionnaire for Paediatric Functional GI Disorders
4. More than 1 loose stool in the 48 hours preceding dosing, that met a Type 6 or Type 7 description on the Bristol Stool Chart
5. Use of any prescription medication, including antibiotics, laxatives and steroids
6. Regular GI complaints, such as stomach upsets, diarrhoea, constipation, flatulence, abdominal colic
7. Known intolerance or sensitivity to any of the study products, abdominal or anorectal surgery
8. Psychiatric disorders, anxiety, and depression
9. Lactose intolerance
10. Use of supplements that may have affected GI system including laxatives, fibre, and iron supplements
11. Exposure to any non-registered drug product within 30 days prior to screening visit.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Difference in the number of participants experiencing at least one stool that met a Type 6 or Type 7 description on the Bristol Stool Chart, within 24 hours after study product intake | within 24 hours after study product intake
  Difference in the number of subjects experiencing at least one stool that met a Type 6 or Type 7 description on the Bristol Stool Chart

SECONDARY OUTCOMES:
Number of subjects who experienced at least one loose or watery stool that met a Type 6 or Type 7 description on the Bristol Stool Chart | in a 24-hour period post-consumption of intervention
  Stool frequency, measured as the number of subjects who experienced at least one loose or watery stool that met a Type 6 or Type 7 description on the Bristol Stool Chart
Frequency of the GI symptom event and frequency of participants reporting GI symptoms events by the severity and causality (i.e., related, not related) for each treatment group recorded at Visits 3, 5 and 7, for pre- and post-dose administration | in the 24-hour period post-consumption
  Report common gastrointestinal symptoms including abdominal pain, bloating, cramping, abdominal rumbling, excess flatus, and and nausea associated with d-allulose consumption. These were reported as the frequency of the event and frequency of participants reporting events by the severity and causality (i.e., related, not related) for each treatment group recorded at Visits 3, 5 and 7, for pre- and post-dose administration. The severity of the event was categorized in three levels (mild, moderate, severe).

IPD SHARING:
Plan to Share IPD: No